CLINICAL TRIAL: NCT04189068
Title: Fatal Cerebral Infarction and Ophthalmic Artery Occlusion After Nasal Augmentation With Hyaluronic Acid - A Case Report and Review
Brief Title: Fatal Cerebral Infarction After Nasal Augmentation With Hyaluronic Acid
Status: Completed | Type: Observational
Sponsor: Xijing Hospital (Other)
Responsible Party: Principal Investigator, Yang Qing, Director Clinical research, Xijing Hospital
Other Study IDs: ky20192199-c-1
Record Dates: First submitted 2019-10-30; First posted 2019-12-06 (Actual); Last update posted 2019-12-06 (Actual); Status verified 2019-12

CONDITIONS: Magnetic Resonance Angiography
Keywords: Cerebral Infarction Hyaluronic Acid Embolism

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
this study discussed the pathogenesis, treatment, and prognosis of severe cerebral infarction and ophthalmic artery occlusion for Aisan induced by hyalruonic acid filler injection.

DETAILED DESCRIPTION:
Intra-arterial thrombolysis and retrobulbar injection of hyaluronidase have been used for HA-induced ophthalmic artery obstruction.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of cerebral infarction

Exclusion Criteria:

* fat embolism

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patient with severe cerebral infarction and ophthalmic artery occlusion after nasal augmentation by HA.
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2019-09-24 (Actual); Primary Completion 2019-10-10 (Actual); Study Completion 2019-10-22 (Actual)

PRIMARY OUTCOMES:
pulse | 0-6 day
  Monitore the "beats per minute over the past 6 days.
blood pressure | 0-6 day
  Monitor the blood pressure and record with mm Hg over the past 6 days.

CONTACTS AND LOCATIONS:
Overall Officials: Ma, Study Director — Xijing Hospital
Locations (1):
- Qing, Xi'an, Shaan XI Province, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Li KT, Huang YH, Chen CH, Chou LW. Delayed-onset cerebral infarction after cosmetic facial injection using hyaluronic acid. J Formos Med Assoc. 2016 Jul;115(7):587-8. doi: 10.1016/j.jfma.2015.11.012. Epub 2016 Jan 4. No abstract available. PMID 26763725